CLINICAL TRIAL: NCT01486511
Title: Pulmonary Embolism After Liver Resection: A Prospective Analysis of Risk Factors
Brief Title: Pulmonary Embolism After Liver Resection
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beaujon Hospital (Other)
Responsible Party: Principal Investigator, Emmanuel Melloul, Medical Doctor, Surgeon, Beaujon Hospital
Other Study IDs: Beaujon
Record Dates: First submitted 2011-12-04; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Liver Disease; Pulmonary Embolism; Thrombophilia; Death
Keywords: Liver disease; Pulmonary embolism; Thrombophilia; Death
MeSH Terms: conditions — Liver Diseases; Pulmonary Embolism; Thrombophilia; Death | interventions — Hepatectomy; 4-((1,4,8,11-tetraazacyclotetradec-1-yl)methyl)benzoic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Liver resection patients: All patients that underwent elective liver resection for both malignant and benign diseases.
  Interventions: Procedure: Liver resection; Radiation: Computed Tomography

INTERVENTIONS:
Procedure: Liver resection — Hepatectomy including both minor and major.
  Other Names: Hepatectomy, liver resection
Radiation: Computed Tomography — Computed Tomography +/- pulmonary angiography
  Other Names: CT, CTPA, CT-PA, MSCT, MSCT-PA

SUMMARY:
Major surgery is associated with a postoperative hypercoagulable state related to the surgical trauma that may lead to thromboembolic complications. To the investigators knowledge, only two series have reported the risk of PE after liver surgery with an incidence of up to 6.3% The purpose of this study is to identify the independent risk factors associated with the development of PE after elective liver surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Malignant liver diseases
* Benign liver diseases

Exclusion Criteria:

* Age <18 years
* Previous history of thromboembolic events
* Living Donor hepatectomies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients that will undergo liver resection for any type of liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary embolism | up to January 2012
  Blood clots in the lungs that may lead to sudden death.

SECONDARY OUTCOMES:
Complications | up to January 2012
  Any type of post-operative complications graded according to the Clavien-Dindo Classification of Surgical Complications
Length of hospital stay | up to January 2012
  The duration of hospitalization in days.
Mortality | up to January 2012
  Post-operative 90-Day Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Belghiti, MD, Principal Investigator — Beaujon Hospital
Locations (1):
- Prof. Jacques Belghiti, Paris, Clichy, France